CLINICAL TRIAL: NCT05855031
Title: The Liver Care Trial: Screening for Liver Disease in Individuals Attending Treatment for Alcohol Use Disorder - a Randomized Controlled Study
Brief Title: The Liver Care Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Novavi (Unknown); Aarhus University Hospital (Other); Frederiksberg University Hospital (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: SJ-995
Record Dates: First submitted 2023-04-20; First posted 2023-05-11 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Alcoholic Liver Disease; Alcohol Use Disorder; Alcohol Abuse; Alcoholism; Fibrosis, Liver; Alcohol-Related Disorders
Keywords: Screening; Fibroscan; Liver stiffness measurement; abstinence
MeSH Terms: conditions — Liver Diseases, Alcoholic; Alcoholism; Liver Cirrhosis; Alcohol-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized concealed allocation to intervention or control
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): An invitation to a liver stiffness measurement (Transient Elastography), to blood sampling and a leaflet on alcohol-related disease.
  Interventions: Diagnostic Test: Transient Elastography
- Control (No Intervention): An invitation to screening by blood sampling with Fib-4

INTERVENTIONS:
Diagnostic Test: Transient Elastography — One transient elastography 1-2 weeks after randomization
  Other Names: Fibroscan; Liver stiffness measurement
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of screening for liver disease with liver stiffness measurement on abstinence or light consumption after 6 months in individuals who are receiving treatment for alcohol use disorder and without a history of liver disease. The investigators will conduct a randomized controlled trial with concealed allocation comparing A) an invitation to a liver stiffness measurement, blood sampling and leaflet on alcohol-related disease (intervention) with B) an invitation to blood sampling (control). The primary outcome is 'abstinence or light consumption' (≤ 10 units/week) throughout the last months, and assessed 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Attending outpatient treatment for alcohol use disorder (international classification of disease version 10: F102: alcohol dependence or F101: harmful alcohol use) at Novavi Køge or Novavi Roskilde
* Informed written consent

Exclusion Criteria:

* Not speaking Danish or English
* Severe liver disease (known by the participant)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol abstinence or light consumption (≤ 10 units/week) the last 30 days (yes/no) assessed 6 months since randomization | Assessed 6 months after randomization
  Assessed By telephone interview or health record

SECONDARY OUTCOMES:
Heavy drinking days last 30 days | Assessed 6 months after since randomization
  Assessed by telephone interview or health record
Change in AUDIT-C score (yes or no) since randomization | 6 months after randomization
  AUDIT: the Alcohol Use Disorders Identification Test is a validated manual for use in primary care to identify persons with hazardous and harmful patterns of alcohol consumption

OTHER OUTCOMES:
Improvement or no decrease in motivation to cut down on alcohol (yes or no) | 6 months after randomization
  Assessed by telephone interview via questionnaire
Improvement or no decrease in physical and mental health-related quality of life (SF-12) (yes or no), calculated as the difference between baseline and follow-up. | Assessed 6 months after randomization
  SF 12 (12-Item Short Form Survey) is a validated self-reported outcome measure assessing the impact of health on an individual's everyday life
Comparing abstinence or light consumption last 30 days between those in the intervention group with a screen negative result with those in the control group. | Assessed 6 months after randomization
  Light consumption < 10 units/week
Comparing alcohol consumption amount between those with a positive fibroscan vs. those with a negative fibroscan | Assessed 6 months after randomization
Improvement or no decrease in smoking (yes/no) | Assessed 6 months after randomization
  By logistic regression

CONTACTS AND LOCATIONS:
Overall Officials: Gro Askgaard, PHD, Principal Investigator — Zealand University Hospital
Locations (2):
- Denmark (2):
  - Novavi Køge, Køge
  - Novavi Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dahlin P, Jepsen P, Molzen L, Madsen LG, Wegmann During S, Benthien KS, Winther-Jensen M, Grew JC, Kirk JW, Jensen KJ, Petersen J, Askgaard G. The Liver Care Trial: screening for liver disease in individuals attending treatment for alcohol use disorder-study protocol for a randomized controlled study. Trials. 2025 Oct 28;26(1):448. doi: 10.1186/s13063-025-09151-8. PMID 41152905

DOCUMENTS (2):
  • Study Protocol (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT05855031/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT05855031/SAP_001.pdf